CLINICAL TRIAL: NCT04262544
Title: An Innovative Mobile Health Intervention to Improve Self-care in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Indiana University (Other); Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Spyros Kitsiou, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-0790; 1R21NR018281-01A1 (NIH)
Record Dates: First submitted 2020-01-06; First posted 2020-02-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
Keywords: mHealth; text messaging; smartphone; mobile apps; wearables; heart failure; self-management; telehealth
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers (doctors and nurses) providing usual care to study participants will be blinded to the allocation of participants.
  Data collectors and assessors of subjective outcomes (e.g. health beliefs, self-efficacy, self-care) will be blinded to the allocation. Study participants will be asked not to reveal to their provider and assessor which group they are assigned to. Data collectors/assessors will have restricted access to patient data in REDCap and will not share the same space with other study investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth (Experimental): Intervention group
  Interventions: Behavioral: iCardia4HF
- Usual Care (Active Comparator): Control group
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: iCardia4HF — Participants in the intervention group will receive the following main components in addition to usual care: 1) the Heart Failure Health Storylines mobile app which supports daily self-monitoring and management of vital signs and symptoms; 2) three connected health devices (Fitbit activity tracker, Withings Cardio Body weight scale and blood pressure monitor), and 3) a program of tailored text-messages targeting health beliefs, self-efficacy, and HF-knowledge.
  Arms: mHealth
Other: Usual Care — Participants assigned to the control group will receive usual care and the same connected health devices (Fitbit activity tracker, Withings weight scale and blood pressure monitor) as patients in the intervention group, but without the heart failure health storylines mobile app and text-messaging program. Usual care includes patient education before hospital discharge, and follow-up visits at the outpatient HF clinic a week after discharge and monthly thereafter depending on the patient's condition. Patient education includes literacy-sensitive, education material about HF self-care developed by the Sheps Center for Health Services Research,and a 40-minute education session with an APN and a dietician to review and discuss the education material provided to the patient.
  Arms: Usual Care

SUMMARY:
Heart failure (HF) is associated with high mortality and hospitalization rates. Prior studies show that adherence to routine HF self-care behaviors reduces the risk of all-cause mortality and HF-related hospitalizations, and improves health related quality of life. However, self-care has generally been found to be poor among HF patients. This study aims to assess the feasibility, acceptance, and efficacy of an innovative, patient-centered intervention (iCardia4HF) that aims to promote adherence to HF self-care and improve patient outcomes through the use of commercially available mobile health technologies.

DETAILED DESCRIPTION:
More than 6.5 million people have heart failure (HF) in the United States and 960,000 new cases are reported annually. HF is associated with high mortality and hospitalization rates, high costs, and poor health-related quality of life (HRQL). Despite major improvements in outcomes with medical and surgical therapy, admission rates following a HF-related hospitalization remain high with 25% of patients readmitted to the hospital within 30-days and up to 50% readmitted within 6 months. Previous research shows that adherence to routine HF self-care behaviors reduces the risk of all-cause mortality and HF-related hospitalization, and improves HRQL. However, self-care has generally been found to be poor among HF patients, particularly minority populations. Nonadherence to HF symptom monitoring and medication use is remarkably high even among recently discharged patients hospitalized due to a HF exacerbation. Recent advances in consumer-based mobile health (mHealth) technologies, such as smartphones, mobile health apps, wearable sensors, and other smart and connected health devices, offer scalable and affordable solutions for promoting better HF self-care and expanding delivery of care services to communities that are difficult to reach. However, no prior studies have assessed the impact of these technologies on HF self-care and patient outcomes.

This study aims to conduct a pilot randomized controlled trial (RCT) of a patient-centered intervention named iCardia4HF that promotes adherence to HF self-care through the use of commercial mHealth devices and app tools. iCardia4HF consists of: (1) a patient-centered mHealth app, developed in partnership with the Heart Failure Society of America, that interfaces with multiple connected health devices and comprises a number of self- monitoring, patient education, and adherence reminder tools for improving self-care; and (2) individually tailored text-messages (TMs) targeting health beliefs, self-care efficacy, and HF-knowledge. Study participants (n=92) diagnosed with HF will be randomly assigned to iCardia4HF or the control group for 12 weeks. Specific aims are to: 1) assess the feasibility and acceptance of iCardia4HF; 2) examine the preliminary efficacy of iCardia4HF on objectively assessed measures of HF self-care using real- time data from the connected health devices and app, as well as self-reported Self-Care and HRQL; track the number of hospitalizations and emergency room (ER) visits over 12 weeks; and 3) examine the mediating effect of intervention target variables (health beliefs, self-care efficacy, and HF-knowledge) and impact of independent patient factors on HF self-care.

This study represents an important step in identifying an affordable and scalable mHealth intervention that has the potential to bring about a new paradigm in self-care management of HF.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HF, Stage C
* ≥ 18 years of age
* Being treated with oral diuretics for heart failure
* Suboptimal HF self-care adherence (score 1 or 2 in at least two items of the Self-care of Heart Failure Index v.7.2)
* Ability to speak and read English

Exclusion Criteria:

* Planned coronary revascularization, Transcatheter Aortic Valve Implantation (TAVI), Cardiac Resynchronization Therapy (CRT) - implantation, and/or heart transplantation (HTx) within the next 3 months.
* Coronary revascularization and/or CRT-implantation within the last 30 days
* Advanced renal disease (stage IV CKD, GFR<30, or hemodialysis)
* Known alcohol or drug use
* End-stage HF (hospice candidate)
* Active cancer
* Pregnancy
* Not able to take care of self (eat, dress, walk, bath, take medications, or use the toilet)
* Discharged to or already living in a nursing home or other care facility other than home
* Cognitive impairment (MoCA score < 22).
* Prior use of study devices for self-care or participation in a similar trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Medication adherence (dose count) | Weeks 1 to 12
  Percent of prescribed number of doses taken
Medication adherence (dose time) | Weeks 1 to 12
  Percent of doses taken on schedule within 25% of the expected time interval
Adherence to daily self-monitoring of weight | Weeks 1 to 12
  Number of days patients completed at least one measurement between 12 am and 11:59pm

SECONDARY OUTCOMES:
Adherence to daily self-monitoring of blood pressure | Weeks 1 to 12
  Number of days patients completed at least one BP measurement between 12 am and 11:59pm
Adherence to self-monitoring of HF symptoms | Weeks 1 to 12
  Number of days intervention patients used the mobile app to record their HF symptoms
Physical activity - Steps | Weeks 1 to 12
  Number of daily steps (measured with a Fitbit device)
Moderate-to-Vigorous Physical Activity | Weeks 1 to 12
  Number of moderate-to-vigorous physical activity minutes per day (measured with a Fitbit device)
Adherence to low-sodium diet | Baseline, 12 Weeks
  Sodium intake will be assessed with a urinary sample test
Self-reported Self-care | Baseline, 30 days, and 12 Weeks
  Measured with the Self-Care Heart Failure Index (SCHFI) v.7.2. Each scale score ranges from 0 to 100. Higher scores indicate better self-care.
Health Beliefs about Medication Compliance | Baseline, 30 days, and 12 Weeks
  Beliefs about Medication Compliance Scale (12-items)
Health Beliefs about Dietary Compliance | Baseline, 30 days, and 12 Weeks
  Beliefs about Dietary Compliance Scale (12 items)
Health Beliefs about Self-Monitoring Compliance | Baseline, 30 days, and 12 Weeks
  Beliefs about Self-Monitoring Scale (18 items)
HF-knowledge | Baseline, 30 days, and 12 Weeks
  HF-specific knowledge will be assessed with the Dutch Heart Failure Knowledge Scale (DHFK), a 15-item questionnaire measuring general knowledge about HF, symptom recognition, and treatment (e.g. diet and fluid restriction)
Health-related Quality of life (HRQoL) | Baseline, 30 days, and 12 Weeks
  HRQoL will be measured with the Kansas City Cardiomyopathy Questionnaire, which contains 23-items that can be quantified into five subscales: physical limitations, symptoms (frequency, severity, and change over time), quality of life (QoL), social interference, and self-efficacy. Lower scores indicate worse HRQoL.

OTHER OUTCOMES:
HF-related hospitalizations | Weeks 1 to 12
  Number of patients with an event
HF-related hospitalization rate | Weeks 1 to 12
  Number of hospitalizations per person
All-cause hospitalizations | Weeks 1 to 12
  Number of patients with an event
All-cause hospitalization rate | Weeks 1 to 12
  Number of all-cause hospitalizations per person
Emergency room visits | Weeks 1 to 12
  Number of patients with an event
Emergency room visit rate | Weeks 1 to 12
  Number of emergency room visits per person

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kitsiou, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital & Health Sciences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Final research data along with metadata and descriptors will be shared to make sharing meaningful and usable by other researchers. More specifically, we will share both de-identified individual-level data and aggregate data in the form of summary statistics and tables. For the individual-level data, we will develop a data dictionary and documentation guide to maximize the utility of the data and to help qualified researchers understand and properly use the data as needed.
Supporting Information: Study Protocol, CSR
Time Frame: Within 2 years after the final data collection is completed or within one year after the publication of the main outcomes manuscript (whichever comes first), we will share the final, completely de-identified dataset with the research community.

REFERENCES:
- [Derived] Kitsiou S, Gerber BS, Kansal MM, Buchholz SW, Chen J, Ruppar T, Arrington J, Owoyemi A, Leigh J, Pressler SJ. Patient-centered mobile health technology intervention to improve self-care in patients with chronic heart failure: Protocol for a feasibility randomized controlled trial. Contemp Clin Trials. 2021 Jul;106:106433. doi: 10.1016/j.cct.2021.106433. Epub 2021 May 13. PMID 33991686